CLINICAL TRIAL: NCT02467556
Title: Psychological Intervention and Physiotherapy With Medication Improves CRPS Patients Outcome
Acronym: MultiModCRPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Hanna Harno, MD, PhD, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Helsinki University Hospital
Record Dates: First submitted 2015-06-08; First posted 2015-06-10 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2015-06

CONDITIONS: CRPS
Keywords: CRPS; intervention; multimodal
MeSH Terms: interventions — Morphine; Memantine; Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intervention (Other): Open label study with psychological intervention and physiotherapy intervention with medication of morphine, memantine for ten weeks (morphine 30mg tbl per day and memantine up to 40mg tbl per day if tolerated).
  Interventions: Drug: Morphine, memantine; Behavioral: Psychological intervention; Other: Physiotherapy intervention

INTERVENTIONS:
Drug: Morphine, memantine — Morphine up to 30 mg per day orally and memantine up to 40 mg per day orally if tolerated for 10 weeks.
  Other Names: Depolan (morphine), Ebixa (memantine)
Behavioral: Psychological intervention — To help patients shift perspective from pain and CRPS-symptoms, to increase body awareness, to create vivid imagenary, to increase the use of a CRPS hand with mindfulness exposure exercises, to increase flexibility in behavioral repertoire, to explore the fusion of emotions, automatic cognitions and learned responses and to help patients to integrate new skills in their lives.
Other: Physiotherapy intervention — Graded motor imagenary with group and individual weekly sessions with daily practices at home.

SUMMARY:
A ten week open label study intervention to evaluate the outcome for a psychological intervention combined with physiotherapy and medication with memantine-morphine in 10 CRPS patients.

DETAILED DESCRIPTION:
Ten CRPS I patients attended an intervention for 10 weeks. First, the medication was started with morphine 10mg adding gradually to 30 mg per day. Then, in addition to morphine, memantine 5 mg was started adding the dose gradually up to 40 mg per day if tolerated. Physiotherapy and psychological intervention were mostly carried out in a weekly group gathering with home exercises that were recorded to a diary. Psychological and physiotherapy interventions lasted for eight weeks. A neurological examination was done before and after the intervention as well as a separate physiotherapist examination of the hands. Patients filled out questionnaires of mood, quality of life, pain, and CRPS descriptions before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* CRPS type 1 for at least 6 months,
* pain NRS 4 or more

Exclusion Criteria:

* major psychiatric or neurological disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Direction of change in patient reported CRPS symptom discriptors | Three months
  Reports of CRPS symptoms

SECONDARY OUTCOMES:
Direction of change in motor parameters | Three months
  Measurements of strength of the hand, the active range of motion in the hand/arm, 9HPT, DASH questionnaire
Direction of change in psychological parameters | Three months
  Patient scores in BDI, PASS-20, CPAQ
Direction of change in quality of life | Three months
  Patient scores in 15D

CONTACTS AND LOCATIONS:
Overall Officials: Eija Kalso, MD, PhD, Study Director — Professor
Locations (1):
- Helsinki University Central Hospital, Helsinki, HUS, Finland

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.

REFERENCES:
- [Background] Bean DJ, Johnson MH, Kydd RR. The outcome of complex regional pain syndrome type 1: a systematic review. J Pain. 2014 Jul;15(7):677-90. doi: 10.1016/j.jpain.2014.01.500. Epub 2014 Feb 12. PMID 24530407
- [Background] Gustin SM, Schwarz A, Birbaumer N, Sines N, Schmidt AC, Veit R, Larbig W, Flor H, Lotze M. NMDA-receptor antagonist and morphine decrease CRPS-pain and cerebral pain representation. Pain. 2010 Oct;151(1):69-76. doi: 10.1016/j.pain.2010.06.022. Epub 2010 Jul 13. PMID 20630656
- [Derived] Elomaa M, Hotta J, de C Williams AC, Forss N, Ayrapaa A, Kalso E, Harno H. Symptom reduction and improved function in chronic CRPS type 1 after 12-week integrated, interdisciplinary therapy. Scand J Pain. 2019 Apr 24;19(2):257-270. doi: 10.1515/sjpain-2018-0098. PMID 30789827